CLINICAL TRIAL: NCT05868070
Title: Feasibility and Safety of In-bed Cycling/Stepping in Critically Ill Patients: A Study Protocol for a Pilot Randomized Controlled Clinical Trial
Brief Title: Feasibility and Safety of In-bed Cycling/Stepping in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyung Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0720234107; 202013C18 (Other Grant/Funding Number: the Korea Medical Device Development Fund)
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Critically Ill Patient; Intensive Care Unit Acquired Weakness
Keywords: clinical trial; critically ill patient; in-bed cycling; in-bed stepping; intensive care unit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The group allocation will be performed by an independent researcher who is not involved in the evaluation of treatment outcomes and be concealed to physiotherapists who are involved in the evaluation of treatment outcomes. The participants and in-bed cycling/stepping intervention provider will be instructed not to disclose the allocation to the evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (No Intervention): Conventional rehabilitation corresponds to general rehabilitation for critically ill patients and is mainly performed according to functional mobility with a range of motion. This includes Lying without contractures, turning self, sitting balance, sitting at the edge, standing and transfer, assisted gait, and gait endurance.
- Conventional rehabilitation plus multimodal exercise (Experimental): Conventional rehabilitation corresponds to general rehabilitation for critically ill patients and is mainly performed according to functional mobility with a range of motion. This includes Lying without contractures, turning self, sitting balance, sitting at the edge, standing and transfer, assisted gait, and gait endurance. Patients in the intervention group additionally receive multimodal exercise using the in-bed cycle/stepper.
  Interventions: Device: Conventional rehabilitation plus multimodal exercise

INTERVENTIONS:
Device: Conventional rehabilitation plus multimodal exercise — Depending on the patient's condition, the intervention gradually progressed to passive, active assistive, active, and resistive exercise modes and the frequency of exercise interventions is gradually increased, and the application time of cycling/stepping is 20 minutes per session, and up to 3 times if there is no serious problem corresponding to the safety standards.
  Arms: Conventional rehabilitation plus multimodal exercise

SUMMARY:
Intensive care unit (ICU)-acquired weakness (ICU-AW) is one of the most common complications of post-ICU syndrome. It is the leading cause of gait disturbance, decreased activities of daily living, and poor health-related quality of life. The early rehabilitation of critically ill patients can reduce the ICU-AW. We designed a protocol to investigate the feasibility and safety of conventional rehabilitation with additional in-bed cycling/stepping in critically ill patients. The study is designed as a single-center, open-label, pilot, randomized, parallel-group study. After the screening, participants are randomly allocated to two groups, stratified by mechanical ventilation status. The intervention group will be provided with exercises of in-bed cycling/stepping according to the level of consciousness, motor power, and function in addition to conventional rehabilitation. In contrast, the control group will be provided with only conventional rehabilitation. The length of the intervention is from ICU admission to discharge, and interventions will be conducted for 20 minutes, a maximum of three times per session. The primary outcome is the number and percentage of completed in-bed cycling/stepping sessions, the duration and percentage of in-bed cycling/stepping sessions, and the number of cessations of in-bed cycling/stepping sessions. The secondary outcomes are the interval from ICU admission to the first session of in-bed cycling/stepping, the number and percentage of completed conventional rehabilitation sessions, the duration and percentage of conventional rehabilitation sessions, the number of cessations of conventional rehabilitation sessions, the number of adverse events, level of consciousness, functional mobility, muscle strength, activities of daily living, and quality of life. This study is a pilot clinical trial to investigate the feasibility and safety of conventional rehabilitation with additional in-bed cycling/stepping in critically ill patients. If the expected results are achieved in this study, the methods of ICU rehabilitation will be enriched.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45
* Admission to ICU ≤ 72 hours
* Patient deemed to need ≥ 48 hours of ICU care
* Premorbid functional ambulation category≥ 2

Exclusion Criteria:

* Neurologic disorders i.Central nervous system: acute stroke, advanced dementia, hypoxic-ischemic encephalopathy ii. Peripheral nervous system: amyotrophic lateral sclerosis, myasthenia gravis, acute inflammatory demyelinating polyneuropathy
* Acute deep venous thrombosis, pulmonary embolism
* Pneumothorax
* External fixator, superficial metallic implants, amputation, eschar, etc
* Expected ICU discharge within 3 days of admission
* Pregnant
* Difficulty in obtaining consent (rejection, no family, if the family does not agree)
* If the life expectancy is less than 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the number and percentage of completed in-bed cycling/stepping sessions | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  the number and percentage of completed in-bed cycling/stepping sessions
the duration and percentage of in-bed cycling/stepping sessions | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  the duration and percentage of in-bed cycling/stepping sessions
the number of cessations of in-bed cycling/stepping sessions | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  the number of cessations of in-bed cycling/stepping sessions

SECONDARY OUTCOMES:
the interval from ICU admission to the first session of in-bed cycling/stepping | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  the interval from ICU admission to the first session of in-bed cycling/stepping
the number and percentage of completed conventional rehabilitation sessions | at every intervention (from baseline to hospital discharge, an average of 2 months)
  the number and percentage of completed conventional rehabilitation sessions
the duration and percentage of conventional rehabilitation sessions | at every intervention (from baseline to hospital discharge, an average of 2 months)
  a 5-item to measure physical function for patients in ICU and consists of 5 the duration and percentage of conventional rehabilitation sessions
the number of cessations of conventional rehabilitation sessions | at every intervention (from baseline to hospital discharge, an average of 2 months)
  the number of cessations of conventional rehabilitation sessions
the number of adverse events | at every intervention (from baseline to hospital discharge, an average of 2 months)
  the number of adverse events
the confusion assessment method for the ICU (CAM-ICU) | baseline-ICU discharge (an average of 3 weeks)
  The CAM-ICU is a short test for the diagnosis of delirium in adult patients in critical care settings. As a tool to evaluate the presence of delirium, it is evaluated by four characteristics. Trait 1 is characterized by acute changes in mental state or fluctuating mental state, trait 2 is characterized by attention deficit, trait 3 is characterized by unsystematic thinking, and trait 4 is characterized by changes in the level of consciousness. The presence of delirium is when the trait 1 and trait 2 are present, and trait 3 or trait 4 is present.
Richmond agitation-sedation scale (RASS) | baseline-ICU discharge (an average of 3 weeks)
  RASS is a valid and reliable assessment tool to measure the level of alertness and agitated behaviour in critically-ill patients.
Functional ambulation category (FAC) | baseline
  FAC is a 6-point functional gait test that assesses walking ability to determine how much support a patient needs when walking, with or without a personal assistive device. Nonfunctional gait is scored as 0, level 2 dependent gait is scored as 1, Level 1 dependent gait is scored as 2, supervised independent gait is scored as 3, independent gait on a flat surface is scored as 4, and independent gait anywhere is scored as 5.
Functional status score (FSS-ICU) | baseline-ICU discharge (an average of 3 weeks)
  a 5-item to measure physical function for patients in ICU and consists of 5 categories: rolling, supine-to-sit transfers, unsupported sitting, sit-to-stand transfers, and ambulation. Each category was rated from 0 to 7, with a maximum cumulative score of 35.
Short physical performance battery score (SPPB) | ICU discharge (an average of 3 weeks)-hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)-3 months after the hospital discharge (an average of 5 months)
  SPPB is a common well-established measurement of physical performance and involves a timed 4-m walk, timed repeated chair sit-to-stand test, and 10-s balance tests including side-by-side, semi-tandem, and full-tandem. Each of the three subtests of the SPPB is scored from 0 to 4, and summed for a total score ranging from 0 to 12.
de Morton Mobility Index (DEMMI) | baseline-ICU discharge (an average of 3 weeks)-hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)
  DEMMI is a 15 item measure of mobility. In bed, three items will be evaluated: bridge, roll onto side, and lying to sitting. In the chair, three items will be evaluated: sit unsupported in chair, sit to stand from chair, and sit to stand without using arms. In the static balance, four items will be evaluated: stand unsupported, stand feet together, stand on toes, and tandem stand with eyes closed. And walking will be evaluated two items: walking distance and walking independence. In the dynamic balance, three items are evaluated pick up pen from floor, walks 4 steps backwards, jump. The DEMMI is considered an important characteristic of independent mobility and includes items that have validity in measuring the mobility domain defined by the World Health Organization. Using a simple conversion table for 15 evaluation items, it can convert ordinal mobility score (out of 19) into interval mobility score (out of 100).
Falls efficacy scale (FES) | hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)-3 months after the hospital discharge (an average of 5 months)
  The FES is a questionnaire that evaluates the fear of falls in daily life at home and is a 16 item questionnaire with a score ranging from minimum 16 to maximum 64.
Activities-specific balance confidence scale (ABC) | hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)-3 months after the hospital discharge (an average of 5 months)
  ABC scale is a valid and reliable instrument to self-reporting measure of evaluates the fear of falling not only inside the house but also outside the house .
Sum of medical research council (MRC) | baseline-ICU discharge (an average of 3 weeks)-hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)
  MRC-sum score is a commonly used for evaluating the strength of the upper and lower extremities from grade 5 to 0. The sum of MRC scores will be evaluated the strength of a total of 12 joints of 6 joints including the arms, elbow, wrist, hip, knee, and ankle on both sides is measured, for a total of 60 points.
Hand grip strength (HGS) | baseline-ICU discharge (an average of 3 weeks)-hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)
  HGS is commonly performed to measure hand muscle power using a dynamometer and provide an objective index of the functional integrity of the upper extremity.
Modified barthel index (MBI) | ICU discharge (an average of 3 weeks)-hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)
  The MBI is a measure of activities of daily living and involves 10 domains of activities including bowel control, bladder control, as well as help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing.
36-Item Short Form Survey (SF-36) version 2.0. | hospital discharge (an average of 2 months)-1 month after the hospital discharge (an average of 3 months)-3 months after the hospital discharge (an average of 5 months)
  SF-36 is a well-researched, self-reported measure of functional health. Each item consists of physical functioning, role limitations physical, bodily pain, general medical health, vitality, social functioning, role limitations emotional, mental health, physical component scale, and mental component scale.
days to initiate ambulation (FAC ≥2) | at every intervention (from baseline to hospital discharge, an average of 2 months)
  days to initiate ambulation (FAC ≥2)
mortality-28 days | at every intervention (from baseline to hospital discharge, an average of 2 months)
  mortality-28 days
duration of mechanical ventilation | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  duration of mechanical ventilation
length of stay in the ICU | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  length of stay in the ICU
length of stay in the hospital | at every intervention (from baseline to hospital discharge, an average of 2 months)
  length of stay in the hospital
Pittsburgh rehabilitation participation scale (PRPS) | at every intervention (from baseline to ICU discharge, an average of 3 weeks)
  PRPS is a clinician-rated instrument designed to assess a patient's participation in therapy. It is evaluated on a scale of 1 to 6 as an evaluation of the patient's effort and activeness participating in treatment.
concomitant occupational therapy and its application dose | at every intervention (from baseline to hospital discharge, an average of 2 months)
  concomitant occupational therapy and its application dose
concomitant pulmonary rehabilitation and its application dose | at every intervention (from baseline to hospital discharge, an average of 2 months)
  concomitant pulmonary rehabilitation and its application dose.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Hyung Lee, MD, PhD, Principal Investigator — Seoul National University Hospital; Soohyun Wi Wi, PhD, Study Director — Seoul National University Hospital; Hyung-Ik Shin, MD, PhD, Study Director — Seoul National University Hospital; Sung Eun Hyun, MD, PhD, Study Director — Seoul National University Hospital; Kwan-Sik Sung, MS, Study Director — Seoul National University Hospital; Jeong Min Kim, MD, Study Director — Seoul National University Hospital; Yae Lim Lee, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wi S, Shin HI, Hyun SE, Sung KS, Lee WH. Feasibility and safety of in-bed cycling/stepping in critically ill patients: A study protocol for a pilot randomized controlled clinical trial. PLoS One. 2024 May 10;19(5):e0301368. doi: 10.1371/journal.pone.0301368. eCollection 2024. PMID 38728323